CLINICAL TRIAL: NCT02974946
Title: Kidney Protection Using the RenalGuard® System in Cardiac Surgery
Acronym: KIDNEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016CAR88
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Acute Renal Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): Patients will receive the RenalGuard system
  Interventions: Device: RenalGuard
- Control group (No Intervention): Standard practice will be performed with no RenalGuard system

INTERVENTIONS:
Device: RenalGuard
  Arms: Study group

SUMMARY:
This is a prospective randomised control trial 1:1 in patients at risk of developing Acute Kidney Injury after cardiac surgery comparing the RenalGuard® System to current medical treatment. 110 patients will be recruited for each group. The aim of the study is to assess whether the RenalGuard® system reduces Acute Kidney Injury (AKI) after cardiac surgery as compared to current practice.

DETAILED DESCRIPTION:
Patients undergoing elective or in-house urgent cardiac surgery will be approached for the KIDNEY study if they fulfil the inclusion criteria. Upon consent pre-operative blood tests will be as per the usual practice. Moreover, 2ml of the serum will be stored for NGAL analysis.

Following the consenting process, patients will be randomised (envelop- based) into either having the RenalGuard® System (Study group) or current medical management (Control group).

Study group:

Patients in the study group will have the RenalGuard® System started in anaesthetic room once the peripheral line and arterial lines are sited. The RenalGuard® System will continue to run throughout the cardiac procedure in the operating room and up to 6 hours post-op after the patient has been transferred to the unit. Patients will be managed at a zero balance i.e. volume of the urine output will be matched to the volume of Hartmann's fluid infusion. Forced diuresis is then initiated.

Control group:

Patients in the control group will be managed as per current medical practice which will include no forced diuresis in operating room and the use of inotropes for maintenance of mean arterial pressure and intravenous furosemide for diuresis.

An additional blood test (NGAL) at six hours post-op will be taken and would require 2mls of blood. The NGAL specimens will be dealt with by the biochemistry lab (centrifuged & stored) so that the specimens can be analysed in batches.

Patients kidney function (U&Es) will be tested at the time of post-operatively as per usual practice (Day1, pre-discharge and as clinically indicated) and at the post-operative surgical out-patient visit.

Pre-operative, intra-operative and post-operative data will be collected for each patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing surgery (elective or in-house urgent)
2. Patient 18 years old and over
3. Patient able to give written consent
4. Patient at risk of developing AKI after cardiac surgery (at least one factor)

   1. Diabetics (IDDM or NIDDM) with normal kidney function pre-op
   2. Patients with eGFR 20-60
   3. Patients undergoing combined cardiac procedures when the CPB time is likely to exceed 120 minutes
   4. Patients with Hb of 12.5 g/dl or below
   5. Logistic Euroscore of 5 and above
5. Patient not involved with another study

Exclusion Criteria:

1. Emergency surgery
2. Patient unable to give written consent
3. Patient already dialysis dependent or eGFR <20
4. Patient partaking in another study
5. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI as defined by the RIFLE criteria | 50% rise in pre-op serum creatinine within 3 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Heyman Luckraz, Principal Investigator — Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

REFERENCES:
- [Result] Luckraz H, Giri R, Wrigley B, Nagarajan K, Senanayake E, Sharman E, Beare L, Nevill A. Reduction in acute kidney injury post cardiac surgery using balanced forced diuresis: a randomized, controlled trial. Eur J Cardiothorac Surg. 2021 Apr 13;59(3):562-569. doi: 10.1093/ejcts/ezaa395. PMID 33236105
- [Result] Luckraz H, Giri R, Wrigley B, Nagarajan K, Senanayake E, Sharman E, Beare L, Nevill A. Balanced forced-diuresis compared to control as a reno-protective approach in cardiac surgery: secondary outcome of a randomized controlled trial, assessment of neutrophil gelatinase-associated lipocalin levels. J Cardiothorac Surg. 2021 Aug 24;16(1):240. doi: 10.1186/s13019-021-01620-w. PMID 34429137
- [Result] Luckraz H, Giri R, Wrigley B, Nagarajan K, Senanayake E, Sharman E, Beare L, Nevill A. Balanced forced-diuresis as a renal protective approach in cardiac surgery: Secondary outcomes of electrolyte changes. J Card Surg. 2021 Nov;36(11):4125-4131. doi: 10.1111/jocs.15925. Epub 2021 Aug 19. PMID 34414606
- [Derived] Luckraz H, Giri R, Wrigley B, Hennessy AM, Nicholas J, Nevill A. The use of the RenalGuard system in cardiac surgery with cardiopulmonary bypass: a first in man prospective, observational, feasibility pilot study. Open Heart. 2017 Oct 10;4(2):e000669. doi: 10.1136/openhrt-2017-000669. eCollection 2017. PMID 29071091